CLINICAL TRIAL: NCT03360591
Title: Functional Assessment in TAVI: FAITAVI
Acronym: FAITAVI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Flavio Ribichini, Principal Investigator, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAITAVI
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease; Aortic Valve Stenosis
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physiologically-guided strategy (Experimental): Patients randomized in this group will undergo stenting of coronary lesions showing FFR values ≤0.80 only.
  * Lesions showing positive FFR measurements (<0.80) must be treated with PCI, before or after TAVI.
  * Lesions showing clearly negative values (FFR >0.80) will not be treated with PCI before TAVI, and repeated FFR and iFR measurements after TAVI are strongly recommended.
  * Lesions showing "borderline" FFR measurements before TAVI (FFR 0.80-0.83), should be measured again (both FFR and iFR) after TAVI, and the decision of treating of deferring treatment in a given lesion will be based on the FFR value obtained after TAVI.
  * In all cases iFR values will be recorded for a post hoc analysis and for validation of the study endpoints according to iFR values.
  Interventions: Device: Physiologically-guided strategy
- Angiographically-guided strategy (Other): Patients allocated in this group will undergo stenting of all coronary stenosis ≥50% as assessed by visual estimation in vessels ≥2.5mm. PCI can be performed before in a previous procedure, or after TAVI, but always within one month, ± 5 days of the valve implantation.PCI in the group randomized to the angio-guided procedure can be performed therefore, either before or after valve implantation, in the same or in different procedures. Implantation of second-generation drug eluting stents (DES) in all interventions is advised, but not mandatory, and the brand of the stent is left to the operators and center's choice.
  Interventions: Device: Physiologically-guided strategy

INTERVENTIONS:
Device: Physiologically-guided strategy — The Angiographically-guided strategy is that of aiming the most complete degree of revascularization based on angiographic evaluation (stenting all coronary stenosis of major branches >2.5mm, with a % coronary stenosis>50% as evaluated by visual estimation.
  The Physiologically-guided strategy is that of treating only lesions with FFR ≤0.80, and leaving on optimal medical treatment lesions with FFR >0.80. The iFR values will be recorded in all patients, and verified in the core laboratory to allow a post-hoc analysis correlating the 0.80 FFR cut-off with different iFR cut-off values, and using the same study end-points.
  Particular attention will be dedicated to the eventual occurrence of clinical events in patients deferred on the bases of FFR values >0.80 that show a discrepancy with positive (<0.89) iFR values to investigate the reliability of the FFR in the aortic stenosis setting. Both groups will receive the same TAVI strategy and optimal medical therapy
  Other Names: Angiographically-guided strategy

SUMMARY:
The aim of this study is to compare the clinical outcome of patients with severe aortic valve stenosis and associated significant coronary artery disease treated with TAVI and a percutaneous myocardial revascularization dictated according to two different strategies:

1. the Angiographically-guided strategy;
2. the Physiologically-guided strategy.

DETAILED DESCRIPTION:
Nowadays there are no clear recommendations about treatment of coronary in patients with severe aortic valve stenosis eligible for percutaneous valve replacement, and those available rely on a "common sense", class C, level of evidence. No randomized trials debride the skein about the best strategy of revascularization in this complex group of patients. In particular, it remains unclear whether it is preferable a preventive treatment or an ischemia-driven revascularization and, in addition, if it is safer and better for patient's health a simultaneous or a staged strategy.

The aim of this study is to compare the clinical outcome of patients with severe aortic valve stenosis and associated significant coronary artery disease treated with TAVI and a percutaneous myocardial revascularization dictated according to two different strategies.

The Angiographically-guided strategy is that of aiming the most complete degree of revascularization based on angiographic evaluation (stenting all coronary stenosis of major branches >2.5mm, with a %DS>50% as evaluated by visual estimation).

The Physiologically-guided strategy is that of treating only lesions with FFR ≤0.80, and leaving on optimal medical treatment lesions with FFR >0.80. The iFR values will be recorded in all patients, and verified in the core laboratory to allow a post-hoc analysis correlating the 0.80 FFR cut-off with different iFR cut-off values, according to recent observations and using the same study end-points.

Particular attention will be dedicated to the eventual occurrence of clinical events in patients deferred on the bases of FFR values >0.80 that show a discrepancy with positive (<0.89) iFR values to investigate the reliability of the FFR in the Aortic Stenosis setting.

Both groups will receive the same TAVI strategy and optimal medical therapy. The study is designed as randomized, prospective, multi.center, open label, experimental trial with medical device. After discharge patients will be contacted at 30 days, 6 - 12 and 24 months after the procedure to assess the general clinical status and at 12 months to assess the occurrence of events included in the primary and secondary endpoints. The duration of study participation is 24 months for enrolment, ad 24 months for final follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Written informed consent
3. Diagnosis of severe native aortic valve disease with the indication to endovascular valve replacement given by Heart Team
4. Diagnosis of at least one coronary stenosis >50% at angiography
5. No specific pharmacologic treatment is required to enter the study

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy
3. Lack of informed consent
4. Impaired left ventricular function
5. Signs or symptoms of acute (unstable) myocardial ischemia
6. Contraindication to adenosine administration (e.g., asthma, chronic obstructive pulmonary disease, heart rate <50 beats/min, and systolic blood pressure <90 mmHg)
7. Reduced survival expectancy due to severe co-morbidities (<1 year)
8. Impossibility to obtain follow-up information
9. The lack of any of inclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2017-11-24 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of the treatment | 12 months
  Composite of all-cause death, myocardial infarction, stroke, major bleeding, need for target vessel revascularization as adjudicated by the Clinical Event Committee

SECONDARY OUTCOMES:
Safety endpoint | 30 days
  Composite of all cause mortality, all strokes (disabling and not disabling), life threatening bleeding, AKI (stages 2 or 3, including need for dialysis), coronary artery obstruction requiring intervention, major vascular complication, valve related dysfunction requiring repeat procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ribichini FL, Scarsini R, Pesarini G, Fabris T, Barbierato M, D'Amico G, Zanchettin C, Gregori D, Lorenzoni G, Piva T, Nicolini E, Gandolfo C, La Spina K, Fineschi M, Gallo F, Baccani B, Petronio AS, De Carlo M, Berti S, Drago A, Saia F, Sclafani R, Esposito G, D'Ascenzo F, Tarantini G; FAITAVI Trial investigators. Physiology vs angiography-guided percutaneous coronary intervention in transcatheter aortic valve implantation: the FAITAVI trial. Eur Heart J. 2025 Dec 19:ehaf974. doi: 10.1093/eurheartj/ehaf974. Online ahead of print. PMID 41417623
- [Derived] Ribichini F, Pesarini G, Fabris T, Lunardi M, Barbierato M, D'Amico G, Zanchettin C, Gregori D, Piva T, Nicolini E, Gandolfo C, Fineschi M, Petronio AS, Berti S, Caprioglio F, Saia F, Sclafani R, Esposito G, D'Ascenzo F, Tarantini G. A randomised multicentre study of angiography- versus physiologyguided percutaneous coronary intervention in patients with coronary artery disease undergoing TAVI: design and rationale of the FAITAVI trial. EuroIntervention. 2024 Apr 15;20(8):e504-e510. doi: 10.4244/EIJ-D-23-00679. PMID 38629420